CLINICAL TRIAL: NCT05058144
Title: Randomised, Placebo-controlled and Acute Study to Investigate the Metabolism of a Novel Alpha-Glucan in Adults
Brief Title: Novel Alpha-Glucan Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20.23.NR
Record Dates: First submitted 2021-06-24; First posted 2021-09-27 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: 3X3
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- novel alpha glucan (Experimental): 50g novel alpha glucan dissolved in 300ml water
  Interventions: Dietary Supplement: Drinkable solution
- glucose syrup (Active Comparator): 50g dissolved in 300ml water
  Interventions: Dietary Supplement: Drinkable solution
- Inulin (Active Comparator): 15g Inulin dissolved in 300ml water
  Interventions: Dietary Supplement: Drinkable solution

INTERVENTIONS:
Dietary Supplement: Drinkable solution — the volunteer will consume the volume 300 ml of water with

SUMMARY:
These are the characteristics of the project:

Monocentric:

Double blind randomized and crossover: you will test all the 3 products in random order.

DETAILED DESCRIPTION:
This study will be randomized, double blind, placebo-controlled, single-center, and 3x3 crossover in design. Eligible participants will be randomized to receive the below products in single dose and in different random sequence, as determined by the randomization system

1. 50 g novel alpha glucan
2. 50 g (rapidly digestible control)
3. 15 g (dietary fiber)

ELIGIBILITY:
Inclusion Criteria:

Healthy status (based on anamnesis) Body mass index (BMI) between 18.5 and 29.9 kg/m2 Able to understand and sign informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women
2. Type I and type 2 diabetes
3. Known food allergy or intolerance to test product
4. Major medical/surgical event in the last 3 months potentially interfering with study procedures and assessments
5. Abnormal bowel transit, history of a gastrointestinal disorder (e.g., inflammatory bowel disease, diverticular diseases, colon cancer), or history of chronic constipation with passage of fewer than 3 spontaneous bowel movements per week on average or chronic or recurrent diarrhea with spontaneous bowel movements more often than 3 times daily
6. Any concomitant medication potentially interfering with study procedures and assessment: such as antibiotics, antiacids, or other medications impacting transit time, colonoscopy, irrigoscopy or other bowel cleansing procedures four weeks prior the test
7. Recent episode of an acute gastrointestinal illness
8. Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer.
9. Smokers
10. Volunteer who cannot be expected to comply with the protocol
11. Family or hierarchical relationships with Clinical Innovation Lab team

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Glucose concentration post ingestion of a test product | 180 minutes
  postprandial glycemic response

SECONDARY OUTCOMES:
insulin response post ingestion of a test product | 180 minutes
  postprandial insulin response
intestinal hydrogen production as measured by breath hydrogen | 240 minutes
  postprandial breath hydrogen

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Innovation Lab, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No